CLINICAL TRIAL: NCT01905527
Title: A Prospective, Parallel Group, Phase IV Study of Three Levels of MS LifeLines ® Support Services Provided to Patients Prescribed Rebif ® for Newly Diagnosed or First-switch Relapsing Remitting Multiple Sclerosis (RRMS)
Brief Title: Adherence Trial With MS LifeLines ® Services
Status: Terminated | Type: Observational
Why Stopped: The study was terminated as per the Sponsor's decision.
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200136-567
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Sclerosis; Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing-Remitting; Rebif; Quintiles Geographic Area Group; Standard Subgroup; Custom Subgroup; RxCrossroads Geographic Area Group
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Standard Services of Group A (Group A1)
  Interventions: Other: Standard Services of Group A (Group A1)
- Customized Services of Group A (Group A2)
  Interventions: Other: Customized Services of Group A (Group A2)
- Group B
  Interventions: Other: Group B

INTERVENTIONS:
Other: Standard Services of Group A (Group A1) — Support services provided in this group will include: Initial field nurse injection training visit; field nurse follow-up and subsequent visits; and follow-up phone calls at periodic intervals
  Groups: Standard Services of Group A (Group A1)
Other: Customized Services of Group A (Group A2) — In addition to the initial field nurse injection training visit and follow-up call, subjects will select from support services including field nurse follow-up visits; follow-up phone calls; email and/or text reminders; subject self-assessment and use of treatment planning tools; and mail/e-mail educational materials.
  Groups: Customized Services of Group A (Group A2)
Other: Group B — Support services provided in this group will include initial field nurse injection training visit and follow-up phone calls at periodic intervals.
  Groups: Group B

SUMMARY:
This is a Phase IV study to compare the current level of MS LifeLines ® (MSLL) services (face-to-face nursing visits and phone contacts) with customized MSLL services, to determine the optimal services to enhance medication adherence and treatment persistence with Rebif ® subcutaneous three times a week.

DETAILED DESCRIPTION:
The proposed study is a web-based, prospective, parallel group, Phase IV, 12-month study of patients receiving support services provided by MSLL and contracted nursing services. Following referral of patients to MSLL, consenting patients will be allocated to one of two groups (2:1), based on their geographic area. Group A will be further randomized 1:1 to the standard services subgroup (Group A1) or a customized services subgroup (Group A2). The standard subgroup will receive phones calls and nurse visits at set intervals. Patients in the custom services subgroup will have the option of selecting as many or as few of the "standard" services they will receive after the initial injection training. Subjects will have the option of receiving educational materials, planning tools, and reminders. Patients allocated to Group B will receive a visit for injection training and the follow-up call and then MSLL phone calls at set intervals. Over a period of 12 months (each month defined as a 28-day period), all subjects will receive support services (nurse visit and follow-up phone call, etc) and complete online assessments (MSRS-R, PDSS, etc).

The primary objective of the trial is to determine the impact of two different levels of support service, group A1 and A2, provided by MSLL within Group A, on adherence to prescribed treatment in newly diagnosed or first-switch relapsing remitting multiple sclerosis (RRMS) subjects.

Secondary Objective:

The secondary objectives are:

* To use a pair wise comparison to determine the impact on adherence of the two different levels of service intervention provided by MSLL not compared in the primary objective (Standard services subgroup of Group A (A1) to Group B and Customized service subgroup of Group A (A2) to Group B)
* To determine the correlation of adherence with subject-reported outcomes and other study data;
* To examine the changes from baseline in subject-reported outcomes in each service arm;
* To examine changes from baseline in risk for non-adherence in each service arm; and
* To determine rate of trial dropout between each service arm

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years at the time of informed consent signature
* Male or female
* Female subjects of child bearing potential who report they are not pregnant at screening and agree to avoid pregnancy during study participation by using adequate contraception, defined as two barrier methods, one barrier method with a spermicide, intrauterine device, or use of oral female contraceptive
* Outpatient status at time of online screening
* Subjects prescribed Rebif by their treating physicians as the first disease-modifying drug (DMD) they have received, or up to one prior treatment with either Rebif, Copaxone ®, Avonex ® , Extavia ®, Betaseron ®, Gilenya™, and Aubagio ® (with accelerated elimination), Tysabri ® and Tecfidera™
* Access to, and ability to use, a computer, a mouse, the internet, and an email address. In addition, subjects in the Group A will be required to have access to a telephone that accepts text messaging (in case randomized to the Custom subgroup)
* Subject-reported ability to complete online assignments and read English
* Electronically verified informed consent before any trial-related activities are carried out

Exclusion Criteria:

* Any combination therapy with another DMD for Multiple Sclerosis (MS) while participating in the trial
* Score of 4 on any of the items of the MSRS-R or a score between 5 and 8, inclusive, on the PDDS
* Surgical intervention planned during the 12-month study period
* Pregnant or breastfeeding. Note subjects who are 90 days postpartum, stable, and do not breastfeed may participate.
* History of malignancy, with the exception of skin cancer completely excised and considered cured;
* History of seizures or unexplained blackouts within 30 days prior to online screening
* Current illegal drug use at the time of online screening;
* Any prior participation in an interventional clinical trial for MS (except for Aubagio ® or Tecfidera™), participation in any trial within 30 days prior to online screening, or current participation in another clinical trial;
* Current treatment of another autoimmune disorder other than stable thyroid disease at the time of online screening
* History of prior treatment for MS with any of the following: alemtuzumab, cyclophosphamide, methotrexate, azathioprine, cyclosporin, intravenous immunoglobulin (IVIg), and plasma exchange
* Other significant subject-reported disease that would exclude the subject from the trial
* Significant renal or hepatic impairment that would compromise completion of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been prescribed to Rebif® treatment by their treating physicians will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Subject-reported adherence to treatment, calculated as percent adherence ([number of actual injections / number of expected injections] * 100), for subjects in the Group A1 compared with subjects in the Group A2 | Month 12

SECONDARY OUTCOMES:
Subject-reported adherence to treatment in Group A1, Group A2 and Group B at Month 12 | Month 12
Subject-reported adherence to treatment in Group A1, Group A2 and Group B at Months 3 and 6 | Months 3 and 6
Subject-reported Multiple Sclerosis Rating Scale- Revised (MSRS-R) in Group A1, Group A2 and Group B | Months 6 and 12
Subject-reported Patient-determined Disease Steps Questionnaire (PDDS) in Group A1, Group A2 and Group B | Months 6 and 12
Subject-reported Multiple Sclerosis Self-management Scale - Revised (MSSM-R) in Group A1, Group A2 and Group B | Months 6 and 12
Subject-reported Multiple Sclerosis International Quality of Life (MusiQoL) in Group A1, Group A2 and Group B | Months 6 and 12
Subject-reported Morisky Medication Adherence Scale-4 (MMAS-4) in Group A1, Group A2 and Group B | Months 2, 6, 9 and 12
Change from Baseline in Subject-reported multiple Sclerosis Rating Scale- Revised (MSRS-R) in Group A1, Group A2 and Group B at Months 6 and 12 | Months 6 and 12
Change from Baseline in Subject-reported Patient-determined Disease Steps Questionnaire (PDDS) in Group A1, Group A2 and Group B at Months 6 and 12 | Months 6 and 12
Change from Baseline in Subject-reported Multiple Sclerosis Self-management Scale - Revised (MSSM-R) in Group A1, Group A2 and Group B at Months 6 and 12 | Months 6 and 12
Change from Baseline in Subject-reported Multiple Sclerosis International Quality of Life (MusiQoL) in Group A1, Group A2 and Group B at Months 6 and 12 | Months 6 and 12
Change from Baseline in Subject-reported score in Morisky Medication Adherence Scale-4 (MMAS-4) in Group A1, Group A2 and Group B at Months 2, 6, 9 and 12 | Months 2, 6, 9 and 12
Percentage of subjects who dropped-out of the trial along with the reasons of dropping out in Group A1, Group A2 and Group B | Month 12
Percentage of subjects with more than 80 percent and 90 percent subject-reported adherence to treatment in Group A1, Group A2 and Group B | Month 12
Percentage of subject demographic characteristics in Group A1, Group A2 and Group B | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Call EMD Serono Medical Information for information on recruiting sites, Boston, Massachusetts, United States